CLINICAL TRIAL: NCT06778538
Title: HPGD Overexpression Attenuates Tumorigenesis and EMT in Clear Cell Renal Cell Carcinoma by Upregulating SLCO2A1
Brief Title: Evaluation of HPGD and SCLO2A1 Expression in Clear Cell Renal Cell Carcinoma Patients
Acronym: HPGD-ccRCC
Status: Completed | Type: Observational
Sponsor: Shang Panfeng (Other)
Collaborators: Lanzhou University Second Hospital (Other)
Responsible Party: Sponsor-Investigator, Shang Panfeng, Professor, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Other Study IDs: 2023A-096
Record Dates: First submitted 2025-01-11; First posted 2025-01-16 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: Clear Cell Renal Cell Carcinoma (ccRCC)
Keywords: HPGD; clear cell renal cell carcinoma; biomarker; prognosis; EMT; tumorigenesis; SLCO2A1
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinogenesis | interventions — Immunohistochemistry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue samples, blood samples, and other relevant biological specimens will be retained for future analysis, including potential DNA extraction for genetic studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Immunohistochemistry; WB; PCR — The intervention will specifically focus on evaluating the role of HPGD in patients with clear cell renal cell carcinoma by classifying them into high-low expression groups based on median HPGD expression values by immunohistochemical scores for prognostic analysis. Protein and RNA were extracted from collected ccRCC tissues for expression verification.

SUMMARY:
This study aims to investigate the role of HPGD in clear cell renal cell carcinoma (ccRCC). Specifically, it will focus on HPGD's impact on proliferation, epithelial-mesenchymal transition (EMT), and prognosis. The study will analyze gene expression data from clinical samples and use techniques like RT-qPCR, Western blotting, and immunohistochemistry to assess HPGD expression levels. Additionally, the research will explore the relationship between HPGD and patient survival outcomes. By elucidating HPGD's contribution to cancer progression, the study seeks to identify potential therapeutic targets for improving renal cancer treatment.

DETAILED DESCRIPTION:
This study is designed to comprehensively explore the role of 15-hydroxyprostaglandin dehydrogenase ( HPGD) in clear cell renal cell carcinoma development and progression. HPGD has been implicated in various cancers, with evidence suggesting its involvement in tumorigenesis, EMT, and poor prognosis. However, its specific function n clear cell renal cell carcinoma (ccRCC) is still unclear. This research will analyze clinical samples, including tumor tissues and normal adjacent tissues, to evaluate HPGD expression through a combination of advanced laboratory techniques such as quantitative real-time PCR (qRT-PCR), Western blotting, immunohistochemistry (IHC) and RNA sequencing.

Furthermore, HPGD-interacting proteins were predicted using STRING and TCGA data, followed by PCR, Western blot validation, and IHC. Mechanistically, HPGD positively correlated with the solute carrier organic anion transporter 2A1 (SLCO2A1), and SLCO2A1 knockdown partially attenuated the tumor-suppressive effects of HPGD overexpression..

This study underscores the tumor-suppressive role of HPGD in ccRCC, highlighting its capacity to hinder cell proliferation and EMT via its interaction with SLCO2A1. Targeting the HPGD-SLCO2A1 axis may offer a promising novel therapeutic approach for ccRCC management.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older. Histologically confirmed diagnosis of clear cell renal cell carcinoma . Measurable disease as per RECIST criteria. Adequate organ function as defined by laboratory tests (e.g., liver, kidney, and hematologic function).

HPGD expression level determined via biopsy or previous analysis. Written informed consent provided.

Exclusion Criteria:

History of other malignancies within the past 5 years, excluding non-melanoma skin cancer or in situ carcinoma.

Prior treatment with HPGD inhibitors or similar targeted therapies. Active or uncontrolled infections. Pregnant or breastfeeding women. Known autoimmune disorders or conditions requiring immunosuppressive therapy. Inability to comply with the study protocol or procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients aged 18 years or older with a confirmed diagnosis of clear cell renal cell carcinoma. Participants will be recruited from oncology clinics and hospitals, and all eligible individuals must have measurable disease as defined by RECIST criteria. Both male and female participants will be included, with no restrictions based on ethnicity or socioeconomic background. Participants will be required to provide informed consent and meet the inclusion criteria related to health status and prior treatments.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
HPGD Expression Levels in clear cell renal cell carcinoma（ccRCC） Patients | 2024.1-2024.6
  The primary outcome will measure the expression levels of HPGD in ccRCC tissues compared to adjacent normal tissues, and its correlation with clinical outcomes such as overall survival (OS) and progression-free survival (PFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Lanzhou University Second Hospital, Lanzhou, Gansu, China

IPD SHARING:
Plan to Share IPD: No
We do not plan to share individual participant data (IPD) with other researchers due to the sensitive nature of the clinical data involved. However, aggregated data and relevant findings from the study will be published in peer-reviewed journals to contribute to the scientific community.

REFERENCES:
- [Background] Monteleone NJ, Moore AE, Iacona JR, Lutz CS, Dixon DA. miR-21-mediated regulation of 15-hydroxyprostaglandin dehydrogenase in colon cancer. Sci Rep. 2019 Apr 1;9(1):5405. doi: 10.1038/s41598-019-41862-2. PMID 30931980
- [Background] Arima K, Komohara Y, Bu L, Tsukamoto M, Itoyama R, Miyake K, Uchihara T, Ogata Y, Nakagawa S, Okabe H, Imai K, Hashimoto D, Chikamoto A, Yamashita YI, Baba H, Ishimoto T. Downregulation of 15-hydroxyprostaglandin dehydrogenase by interleukin-1beta from activated macrophages leads to poor prognosis in pancreatic cancer. Cancer Sci. 2018 Feb;109(2):462-470. doi: 10.1111/cas.13467. Epub 2018 Jan 27. PMID 29224225
- [Background] Myung SJ, Rerko RM, Yan M, Platzer P, Guda K, Dotson A, Lawrence E, Dannenberg AJ, Lovgren AK, Luo G, Pretlow TP, Newman RA, Willis J, Dawson D, Markowitz SD. 15-Hydroxyprostaglandin dehydrogenase is an in vivo suppressor of colon tumorigenesis. Proc Natl Acad Sci U S A. 2006 Aug 8;103(32):12098-102. doi: 10.1073/pnas.0603235103. Epub 2006 Jul 31. PMID 16880406
- [Background] Wolf I, O'Kelly J, Rubinek T, Tong M, Nguyen A, Lin BT, Tai HH, Karlan BY, Koeffler HP. 15-hydroxyprostaglandin dehydrogenase is a tumor suppressor of human breast cancer. Cancer Res. 2006 Aug 1;66(15):7818-23. doi: 10.1158/0008-5472.CAN-05-4368. PMID 16885386